CLINICAL TRIAL: NCT02812277
Title: Retrospective Analysis of Effectiveness and Safety Profile of Anastrozole and Letrozole in Adjuvant Treatment of HR+ Early Breast Cancer Patients
Brief Title: Retrospective Analysis of Effectiveness and Safety Profile of Anastrozole and Letrozole in HR+ Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2015014
Record Dates: First submitted 2016-05-15; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: anastrozole; letrozole; postmenopausal patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anastrozole treatment group: The study group was about HR positive postmenopausal breast cancer patients who were hospitalized between January, 2008 and October, 2010, and ever accepted anastrozole therapy with the completed follow-up data.
- letrozole treatment group: The study group was about HR positive postmenopausal breast cancer patients who were hospitalized between January, 2008 and October, 2010, and ever accepted letrozole therapy with the completed follow-up data.

INTERVENTIONS:
Other:  — This is a Non-Interventional Study, so there are no drug or devices included.

SUMMARY:
This is a single centre, observational and retrospective clinical study. The study group was about all HR positive postmenopausal breast cancer patients who were hospitalized between January, 2008 and October, 2010, and ever accepted AI therapy with the completed follow-up data.

DETAILED DESCRIPTION:
The department of surgery at Tian Jin Medical University Cancer Hospital, one of the centers of excellence to treat patients with breast cancer in China, collects and maintains an electronic database of patients treatment details and follow up data. This is a single centre, observational and retrospective clinical study. The study group was about all HR positive postmenopausal breast cancer patients who were hospitalized between January, 2008 and October, 2010, and ever accepted AI therapy with the completed follow-up data.All the enrolled patients received breast-conserving surgery or whole breast surgery, and afterwards, received adjuvant chemotherapy according the pathological types. The patient's clinical pathological data include the age, family history, surgery options, pathologic type, the size of tumor, lymph node status, histological grade, chemotherapy regime, irradiation regime, and the expressions pattern of Her-2 and Ki-67. The research starts when the patients received the first time AI treatment. In the subsequent treatment, we analyzed the patients' bone density changes (T value >-1 indicates normal,-2.5≤T value≤-1 indicates mild osteoporosis, T value <-2.5 indicates severe osteoporosis) each half year for 3 years, analyzed the patients' liver function and kidney function changes each half year for 3 years (AST, ALT, ALP, TBIL, DBIL,UREA and CREA values > 2 times ULN indicates abnormal), analyzed the patients' blood-lipoids (LDL, HDL, TG and TC) each half year for 3 years, the occurrence rates of adverse reactions (skin flush, joint pain, headache, rash, nausea, vomiting, diarrhea, et al), the causes and rates of treatment termination between the 2 groups, the 3 years DFS and OS between two groups, and the factors associated with survival and prognosis, and identified the benefit individuals of AI therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1). Breast cancer confirmed by histology or cytology with the tumor complete resection 2). ER and /or PR positive 3). Postmenopausal woman, defined as a woman fulfilling any 1 of the following criteria (based on the NCCN definition of menopause [National Comprehensive Cancer Network 2008]):

  1. Prior bilateral oophorectomy;
  2. Age ≥ 60 years;
  3. Age < 60 years and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and plasma FSH and estradiol in the postmenopausal range; if taking tamoxifen or toremifene, and age<60 years, then serial measurement of plasma FSH and estradiol are need to ensure in the postmenopausal ranges.

     4). Patients have received regular anastrozole or letrozole adjuvant treatment 6). The values of AST, ALT, ALP, TBIL, UREA, CREA were less than 2 times of ULN at the beginning of AI therapy.

     7). BMD T >-1 at baseline.

     Exclusion Criteria:
* Any of the following is regarded as a criterion for exclusion from the study:

  1. . Previous use of the other AIs except for anastrozole or letrozole
  2. . Any severe concomitant condition before AI treatment: uncontrolled cardiac disease or uncontrolled diabetes mellitus et al.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single centre, observational and retrospective clinical study.The study group was about all HR positive postmenopausal breast cancer patients,and ever accepted AI therapy with the completed follow-up data. The patient's clinical pathological data include the age, family history, surgery options, pathologic type,et al. We analyzed the patients' bone density changes, liver function and kidney function changes,and analyzed the patients' blood-lipoids each half year for 3 years, the occurrence rates of adverse reactions, the causes and rates of treatment termination between the 2 groups, the 3 years DFS and OS between two groups, and the factors associated with survival and prognosis, and identified the benefit individuals of AI therapy.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Compare the proportion of patients with abnormal biochemical test results including liver function, kidney function, blood-lipoids, bone density index. | one year

SECONDARY OUTCOMES:
To explore the proportion of patients discontinue AI treatment and reasons related to these discontinuation. | one year
To explore the 3-year DFS rate among the people under upfront therapy. | one year
To explore the 3-year OS rate among the people under upfront therapy. | one year
To explore the DFS in the patients who quit treating. | one year
To explore the OS in the patients who quit treating. | one year

IPD SHARING:
Plan to Share IPD: No